CLINICAL TRIAL: NCT05614505
Title: Efficacy and Acceptability of Ready-to-use Therapeutic Foods (RUTFs) in Indonesia
Brief Title: Efficacy and Acceptability of RUTFs in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Savica (Unknown); UNICEF (Other)
Responsible Party: Principal Investigator, Frank Wieringa, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RUTF_2021_Impact
Record Dates: First submitted 2021-09-22; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Severe Acute Malnutrition
Keywords: Ready to use therapeutic food (RUTF); acceptability; local; children; rehabilitation
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Given the very different characteristics of the RUTFs, full masking is not possible. Caregivers/mothers are only given 1 product, and do not know of the existence of the other intervention products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RUTF standard (Active Comparator): PlumpyNut
  Interventions: Dietary Supplement: Ready to use therapeutic foods
- RUTF local_1 (Experimental): Soybean RUTF
  Interventions: Dietary Supplement: Ready to use therapeutic foods
- RUTF local_2 (Experimental): Mungbean-thick RUTF
  Interventions: Dietary Supplement: Ready to use therapeutic foods
- RUTF local_3 (Experimental): Mungbean-thin RUTF
  Interventions: Dietary Supplement: Ready to use therapeutic foods
- RUTF local_4 (Experimental): Wafer RUTF
  Interventions: Dietary Supplement: Ready to use therapeutic foods

INTERVENTIONS:
Dietary Supplement: Ready to use therapeutic foods — locally produced therapeutic foods

SUMMARY:
Severe wasting or Severe Acute Malnutrition (SAM) continues to be a major public health problem in Indonesia, affecting more than 2 million children under 5 years old. A new approach to treat SAM is called Community-based management of acute malnutrition (CMAM), which has been designed to maximize the coverage and successful treatment of children with SAM, by providing Ready to Use Therapeutic Food (RUTF) through out-patient treatment. Since 2019, UNICEF has been working intensively to facilitate the local production of RUTF. This present study aims to assess the acceptability and efficacy of three locally produced RUTFs compared to the standard peanut based RUTF.

The study will be implemented in Bogor district. A total of 300 children with uncomplicated SAM, aged 6-59 months old, meeting the inclusion criteria will be included in the study. This study is designed as a randomized controlled trial. The children will be allocated to one of the five intervention (1 control, 4 experimental) arms. Each child will receive one type of RUTF product for eight consecutive weeks. The ration given to a child will be based on the need for an intake of ~ 170 kcal/kg BW/day. Data will be collected at baseline, at weekly intervals and at exit. The primary outcome of interest for the efficacy study is the relative weight gain of children consuming each of the local RUTFs compared with those consuming the standard RUTF. The primary outcome of the acceptability of the RUTFs will be the amount of product consumed during the eight-week efficacy trial.

Differences in weight and height gain will be analyzed using ANCOVA, controlling for age, gender, food intake, and morbidity. Repeated measurement statistics will be used to analyze differences in growth patterns over the eight-week intervention.

DETAILED DESCRIPTION:
OBJECTIVES This study aims to assess the acceptability and efficacy to increase weight and mid upper arm circumference of children aged 6-59 months with severe acute malnutrition (SAM), of three locally produced RUTFs compared to the standard peanut based RUTF. The study will be implemented in Bogor district.

METHODOLOGY Subjects inclusion criteria are reported elsewhere.

Sample Size Calculation If the Indonesian RUTFs fulfil the WHO requirement of an average increase of 4 g/kg BW/day, a sample size of 60 children per group would allow detecting a 20% difference between control and intervention products, assuming a SD of 1.6 g/kg BW, a study design effect of 1.0, a significance of 0.05, a power of 0.80. If children fail to reach this 4 g/kg BW target and only gain 2 g/kg BW/day, the sample size would still allow detection of a 30% difference between the control product and the local product. Since it will be a five-armed intervention, a total of 300 SAM children will be recruited in Bogor district.

Anthropometric and Hemoglobin Measurements Training The training on anthropometric measurements will include repeated practice and comparison of intra- and inter-observer variation to ensure that the field team will have excellent skills in conducting the anthropometric measurements.

Hemoglobin concentration will be measured using Hemocue 201+ device by (or under direct supervision of) a medical doctor, trained in the use of the equipment.

Study Design This study is designed as an individually randomised controlled trial. Parents will be informed of the purpose, risks and benefits of the study and asked to sign the informed consent prior to inclusion of their child in the study.

Each child will be randomly allocated to one of the five intervention arms.

Acceptability Study The primary outcome of the acceptability of the RUTFs will be the amount of product consumed during the 8-week efficacy trial (long-term acceptability). An average consumption of at least 50% of the offered product during the 8-week efficacy trial will be considered acceptable.

The secondary outcome of the acceptability study will be the consumption velocity of the RUTFs during the appetite test (short-term acceptability; see below).

Efficacy Study The primary outcome of interest for the efficacy study is the relative weight gain of children consuming each of the local RUTFs compared with those consuming the standard RUTF. A difference of 20% in weight gain will be considered as physiologically significant.

Randomization Prior to the appetite test, selected children with uncomplicated SAM will be randomized to one of the five intervention arms. The randomization list is made prior to recruitment by a member of the research team not present in the field (FTW). Children randomized to one arm will receive the standard RUTF product, and the other four arms will each receive one of four local RUTFs.

Appetite Test The day after the screening, selected children will need to pass an appetite test prior to enrolment in the intervention.

Design Each child will receive one type of RUTF products for eight consecutive weeks. Data will be collected at baseline, at weekly intervals and at exit. Children who completely refuse to eat the RUTF they have been allocated to for more than 4 days/week, for 2 consecutive weeks, or children who lose or do not gain weight during 2 consecutive weekly visits, and/or develop allergic reaction and clinical symptoms during the course of the study will be dropped from the study and will be referred to the Puskesmas for treatment.

A weekly supply of RUTF will be supplied during each of the weekly check-up visits.

Baseline data General information on socio-economic status of the family, ethnicity, educational level of both parents, household food security, IYCF including 24 h food recall, use of micronutrient supplements (vitamin A, iron, syrup) and supplementary foods (PMT/Local PMT), morbidity history and current morbidity, duration of pregnancy, birth weight, immunization status, deworming, sex and age of the child, will be collected at baseline, in addition to height/length, weight, MUAC and hemoglobin concentration. All data will be recorded using a digital questionnaire on tablet computers.

Monitoring The daily amount of RUTF intake of each child will be recorded by the mother/caregiver in a monitoring book provided by the study team. The field team will visit each child on a weekly basis to monitor the feeding and intake recording by the mother/caregiver, as well as any intra-household sharing of the RUTF.

In addition to the weekly home visits, the PL will maintain regular daily communication with the mothers/caregivers through text messages.

Data Analysis The baseline, monitoring, and endline data will be entered in a digital questionnaire by the field workers. The researcher will extract data from digital questionnaire into SPSS format. Data analyses will be done using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Children with uncomplicated SAM (WHZ < -3 and/or MUAC <115 mm) qualified for outpatient treatment, or nutritional edema regardless of anthropometry
* Aged 6-59 months old upon enrolment
* Pass appetite test
* Never received in- and outpatient treatment on SAM (including not having consumed RUTF, F75, F100 or special medical specialty food1 in the last two months
* Willing to participate in the study (parent signed the informed consent)

Exclusion Criteria:

* Body weight < 4.0 kg;
* Uncontrolled or untreatable systemic opportunistic infection, such as active TB, HIV;
* Obvious dysmorphic features, general mental health problems (e.g., Down syndrome, etc.), other conditions interfering with normal growth;
* Participating in another clinical trial;
* Any congenital disorder that interferes with normal nutrient intake; chronic conditions including but not exclusively disorders of heart, kidney or liver (children to be screened by a physician);
* SAM with complications requiring hospital treatment (including edema +3);
* Severe anemia (Hb<7g/dL);
* Is a twin or multiple;
* Allergy to milk, nuts, legumes and/or antibiotics (Amoxicillin and Ampicillin)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
short-term acceptability | consumption of at least 50% of RUTF provided in a 30 minute period
  Passing the appetite test
long-term acceptability | Number of children not finishing the 8 week intervention
  drop-out during the intervention
weight gain over the 8 week intervention | weight gain expressed as weight gain (g)/kg body weight per day over the 8 week intervention
  weight gain (in g) over 8 week intervention

SECONDARY OUTCOMES:
recovery rate | from baseline to end of the 8 week intervention
  percentage of children having WHZ>-2 and/or MUAC >125 mm
increase in height for age Z scores (HAZ) | from baseline to the end of the 8 week intervention
  changes in length growth among the intervention arms
length of stay in the treatment | 8 week intervention or shorter
  Average number of day in treatment to reach recovery or drop-out
Morbidity during the intervention | from baseline to 8 week intervention
  number of sick days based on the weekly recall data
Perception | based on the interview with the caregiver after the 8 week intervention
  Acceptability of the product by caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Frank Wieringa, MD PhD, Principal Investigator — Institute de Recherche pour le Développement
Locations (1):
- Savica, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Yes, IP data will be available upon request